CLINICAL TRIAL: NCT03825445
Title: GnRH Agonist Versus hCG Trigger in Ovulation Induction With Intrauterine Insemination: a Randomized Controlled Trial
Brief Title: GnRH Agonist Versus hCG Trigger in Ovulation Induction With Intrauterine Insemination.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hue University of Medicine and Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H2016/205
Record Dates: First submitted 2019-01-11; First posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Ovulation Induction
Keywords: GnRH agonist trigger; hCG trigger; ovulation induction
MeSH Terms: interventions — Chorionic Gonadotropin

STUDY DESIGN:
Intervention Model Description: A prospective randomized comparative study was conducted at Hue University Hospital in Vietnam. Total of 197 infertile women were randomly assigned to receive either GnRHa trigger (n=98 cycles) or hCG trigger (n= 99 cycles) for ovulation trigger. Patients returned for ultrasound monitoring 24 hours after IUI to confirm ovulation.
Who Masked: Participant, Investigator
Masking Description: Odd even rule
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GnRHa trigger (Experimental): Infertile patients underwent ovarian stimulation, started on cycle day eight with 75 IU Menogon (Ferring Pharm Co, Switzerland) daily. Ultrasound monitoring was required after every 2-3 days of stimulation and adjustments to dose and duration were tailed according the patient's response. Ovulation was triggered when at least one and no more than 3 follicles reached ≥18mm in diameter. Patients were then randomly assigned to receive two doses of GnRH-a (Fertipeptil 0.1mg x 2 vial; Ferring Pharm Co, Switzerland) for ovulation trigger.
  Interventions: Drug: GnRHa (Fertipeptil 0.1mg)
- hCG trigger (Experimental): Infertile patients underwent ovarian stimulation, started on cycle day eight with 75 IU Menogon (Ferring Pharm Co, Switzerland) daily. Ultrasound monitoring was required after every 2-3 days of stimulation and adjustments to dose and duration were tailed according the patient's response. Ovulation was triggered when at least one and no more than 3 follicles reached ≥18mm in diameter. Patients were then randomly assigned to receive hCG (Pregnyl 5000IU; Organon Pharm Co, Nertheland) for ovulation trigger.
  Interventions: Drug: hCG (Pregnyl 5000IU)

INTERVENTIONS:
Drug: GnRHa (Fertipeptil 0.1mg) — Two doses of GnRH-a (Fertipeptil 0.1mg x 2 vial) for ovulation trigger after ovarian stimulation for IUI.
  Arms: GnRHa trigger
Drug: hCG (Pregnyl 5000IU) — hCG (Pregnyl 5000IU) for ovulation trigger after ovarian stimulation for IUI.
  Arms: hCG trigger

SUMMARY:
This study aims to compare clinical pregnancy rates (CPR) in patients who are administered either Gonadotropin-releasing hormone agonists (GnRHa) or human chorionic gonadotropin (hCG) for ovulation trigger in intrauterine insemination (IUI) cycles. A prospective randomized comparative study was conducted at Hue University Hospital in Vietnam. Total of 197 infertile women were randomly assigned to receive either GnRHa trigger (n=98 cycles) or hCG trigger (n= 99 cycles) for ovulation trigger. Patients returned for ultrasound monitoring 24 hours after IUI to confirm ovulation. A clinical pregnancy was defined as the presence of gestational sac with fetal cardiac activity.

DETAILED DESCRIPTION:
Study design A prospective randomized comparative study was conducted at Hue University Hospital in Vietnam from April 2016 to June 2017 in 197 infertile women undergoing IUI. The study was approved by the Ethics Committee at Hue University of Medicine and Pharmacy.

Study population A total of 217 women were recruited into the sample at the first stage. Inclusion criteria were women with bilateral tubal patency, at least one follicle ≥ 18mm in diameter on the day of trigger, and men with more than five millions total motile sperm after preparation. Only the first cycles of IUI were studied and there were 197 infertile women who obtained at least 1 mature follicle at the first cycle were included in analysis. Patients were randomly assigned to receive either GnRHa trigger (n=98 cycles) or hCG trigger (n= 99 cycles) for ovulation trigger.

Intervention All patients included in the study were subjected to complete history and physical. Patients with a history of abnormal menstrual cycles (amenorrhea, oligomenorrhea) underwent ovarian stimulation. Stimulation was started on cycle day eight with 75 IU Menogon (Ferring Pharm Co, Switzerland) daily. Ultrasound monitoring was required after every 2-3 days of stimulation and adjustments to dose and duration were tailed according the patient's response. Ovulation was triggered when at least one and no more than 3 follicles reached ≥18mm in diameter. Patients were then randomly assigned to receive either two doses of GnRH-a (Fertipeptil 0.1mg x 2 vial; Ferring Pharm Co, Switzerland) or hCG (Pregnyl 5000IU; Organon Pharm Co, Nertheland) for ovulation trigger.

IUI was then performed with sperm preparation by radiant centrifugation 36 hours after the trigger. Luteal phase support with progesterone 200mg daily (Utrogestan; Besins Health Care Com, Belgium) was started in the day of IUI.

Assessment of outcomes Patients returned for ultrasound monitoring 24 hours after IUI to confirm ovulation which is determined by the accumulation of free fluid in peritoneum at Douglas sac and disappearance of the previous mature follicles.

Serum β-human chorionic gonadotropin (βhCG) was collected 14 days after insemination. A biochemical pregnancy was defined by βhCG concentration > 25 mIU/ml (Shapphire 350; Cork Com, Ireland). Two weeks after a positive βhCG test, the patient returned for an ultrasound appointment. A clinical pregnancy was defined as the presence of gestational sac with fetal cardiac activity.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women who were indicated for IUI cycles
* bilateral tubal patency
* at least one follicle ≥ 18mm in diameter on the day of trigger, and
* men with more than five millions total motile sperm after preparation.
* Only the first cycles of IUI were studied

Exclusion Criteria:

* No mature follicle
* Disagree to be enrolled

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Infertile women with ovulation stimulation
Enrollment: 197 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
The effectiveness of GnRHa versus hCG in ovulation induction | 14 months
  To compare the ovulation rate of patients who were triggered with GnRHa versus hCG in patients undergoing either natural cycle or controlled ovarian stimulation with gonadotropins and IUI.
The effectiveness of GnRHa versus hCG in pregnancy rate | 14 months
  To compare the pregnancy rate of patients who were triggered with GnRHa versus hCG in patients undergoing either natural cycle or controlled ovarian stimulation with gonadotropins and IUI.

CONTACTS AND LOCATIONS:
Overall Officials: Minh Tam Le, Prof.MD.PhD, Study Director — Hue University of Medicine and Pharmacy, Hue University